CLINICAL TRIAL: NCT04525716
Title: What Are the Effects of the Covid-19 Pandemic Among Operated Patients? A Hospital Based Cohort in Stockholm, Sweden
Brief Title: The Effect of the Covid-19 Pandemic Among Operated Patients
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Andreas Älgå, MD, PhD, Karolinska Institutet
Other Study IDs: CovidKirurgi
Record Dates: First submitted 2020-08-21; First posted 2020-08-25 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Covid19; Surgery
MeSH Terms: conditions — COVID-19 | interventions — Social Class

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID-19: Patients with confirmed COVID-19 infection
  Interventions: Other: COVID-19 infection status
- Non-COVID-19: Patients without confirmed COVID-19 infection
  Interventions: Other: COVID-19 infection status
- Socioeconomic status: Patients with varying socioeconomic status will be compared
  Interventions: Other: Socioeconomic status

INTERVENTIONS:
Other: COVID-19 infection status — The investigators will compare patients with/without confirmed COVID-19 infection
  Groups: COVID-19; Non-COVID-19
Other: Socioeconomic status — Patients from different socioeconomic groups will be compared
  Groups: Socioeconomic status

SUMMARY:
This project covers several research aims and uses different research methods, such as cohort analyses.

DETAILED DESCRIPTION:
Background:

A novel Coronavirus (SARS-CoV-2) was first detected in the Hubei Province in China in December, 2019. The virus causes a severe respiratory disease (Coronavirus disease 2019, COVID-19) that has rapidly spread worldwide. The COVID-19 pandemic is prognosed to affect a majority of the world's population before the end of 2020. Throughout the course of the pandemic, patients will continuously need essential healthcare, such as for acute surgical conditions. How the clinical course and management of surgical conditions is influenced by concomitant COVID-19 is largely unknown. There is an acute need for an improved evidence base to inform treatment strategies and guide the management of this patient group.

Objectives of initial analyses:

1. To compare confirmed COVID-19 patients with non-COVID-19 patients who undergo surgical treatment and study factors associated with good or bad outcomes.

Methods:

The study will enroll consecutive patients that undergo surgical treatment in the Stockholm Region. Data will be extracted from a series of linked electronic systems, such as electronic healthcare records systems, and regional data systems. Collected data will include routine clinical data, such as baseline characteristics, previous medical history, details on care given at the hospital and data from follow-up visits. Endpoints include death, length of hospital stay and complications, such as readmission, reoperation, sepsis, respiratory failure, and number of days in the intensive care unit. Outcome data of patients with confirmed COVID-19 will be compared to those of patients without COVID-19.

Objectives and methods of further analyses:

By comparing surgical patients from different socioeconomic groups the investigators aim to assess whether socioeconomic status is associated with good or bad outcomes.

Dissemination and relevance:

To the best of the investigators knowledge, there has been no previous comprehensive comparative research on patients with and without confirmed COVID-19 that undergo surgical treatment.

The results will be disseminated through peer-reviewed publications, aiming for journals with a rapid editorial process, preferably open access journals. The findings are expected to increase the knowledge to establish best-treatment strategies and improve outcomes, both for patients affected by COVID-19 and by future epidemics.

ELIGIBILITY:
Inclusion Criteria:

* Patients that undergo surgical treatment in the Stockholm Region during the study period

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that undergo surgical treatment in the Stockholm Region during the study period
Sampling Method: Probability Sample
Enrollment: 300000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Death | 30 days post surgery
  Mortality

SECONDARY OUTCOMES:
Length of stay | Through study completion, an average of 1 month
  Length of hospital stay
Complications | 3 months post surgery
  Includes readmission, reoperation, infection, sepsis, respiratory failure, and number of days in the intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Martin Nordberg, MD, PhD, Study Chair — Karolinska Institutet, Södersjukhuset
Locations (1):
- All acute care hospitals in Region Stockholm, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No